CLINICAL TRIAL: NCT02295527
Title: Effectiveness of a Physical Exercise Intervention Program in Improving Functional Mobility in Older Adults After Hip Fracture in Later Stage Rehabilitation: a Randomized Clinical Trial
Brief Title: Functional Later Rehabilitation in Older Adults: Effectiveness of Physical Exercises
Acronym: REATIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Monica Rodrigues Perracini, Professor at Master's and Doctoral Programs in Physical Therapy, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 27398814.7.0000.0064
Record Dates: First submitted 2014-11-03; First posted 2014-11-20 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home-based physical exercise (Experimental): Participants randomized to the Intervention Group (IG) will be submitted to a physical exercise program involving a progressive and challenging balance training and a neuromuscular and functional training of the lower limbs, conducted at home by physiotherapists, once a week, lasting about one hour, in the first, second and third month after randomization and will be oriented to perform exercises, twice a week, through a booklet. Visits to follow up exercises progression will be conducted once a month, from de fourth to the sixth month and each two months until the end of the follow up at the 12th month, summing up 18 sessions. Participants will receive monthly phone calls to increase exercise adherence.
  Interventions: Other: Home-based physical exercise intervention
- Control Group Usual Care (Other): This group will receive usual care and the booklet regarding bone health information.
  Interventions: Other: Control Group Usual Care

INTERVENTIONS:
Other: Home-based physical exercise intervention — Progressive strengthening of muscle groups ankle dorsi flexors, knee extensors and hip abductors and progressive balance training according to individual capacity:weight-bearing, limits of stability, change of position/direction, maintenance of static and dynamic stability, anticipatory adjustments using different bases of support and different sensory conditions. Dynamic exercises involving spin on its own axis, sitting and standing, up and down stairs, functional reach, steps in different directions and walk training. In the first session the physiotherapist will choose two exercises that best address the participant function goals and will add more exercises each week according to the level of participants' ability and motivation. Participants will receive a detailed booklet, containing photos and instructions of the12 exercises.Visits to follow up exercises will be conducted by the physiotherapists to progress the exercises.
  Other Names: REATIVE
  Arms: Home-based physical exercise
Other: Control Group Usual Care — This group will receive usual care and will not have any disadvantage in participating in the study. We understand that usual care is what participant receives based on the network of health care in which he/she is inserted. The participants will receive at baseline assessment a diary falls logbook and a guidance booklet containing information about prevention of falls, fractures and bone health that will be explained at the moment.
  Other Names: Usual care
  Arms: Control Group Usual Care

SUMMARY:
Hip fractures resulting from falls increase substantially with advancing age and less than a half of the elderly that have sustained and survived after the surgery regain their former levels of mobility. There is increasing evidence that rehabilitation interventions involving exercises and extended beyond the sub acute phase or even in a later stage of care have a positive impact on various functional abilities. The purpose of this study is to determine if an exercise program training for people who have suffered a fall-related hip fracture will improve functional mobility when compared with usual care. Randomized controlled trial using blinded assessors and intention-to-treat analysis. We will recruit 82 older adults, 60 years or over who have suffered a hip fracture due to a fall and have or have not completed physiotherapy and/or rehabilitation. These participants will be in a later stage rehabilitation phase (6 months up to 2 years after the fracture). Participants randomized to the Intervention Group (IG) will be submitted to a physical exercise program involving a progressive and challenging balance training and a neuromuscular and functional training of the lower limbs, conducted at home by physiotherapists, once a week, lasting about one hour, in the first, second and third month after randomization and will be oriented to perform exercises, twice a week, through a booklet. Visits to follow up exercises progression will be conducted once a month, from de fourth to the sixth month and each two months until the end of the follow up at the 12th month, summing up 18 sessions. Participants will receive monthly phone calls to increase exercise adherence. The control group will receive usual care. The primary outcome will be mobility-related disability and participants will be assessed in the baseline, at the end of the intervention (3 months), at 6 and 12 months. The participants will receive monthly phone calls to investigate falls and exercise adherence. Adverse effects will be monitored.

DETAILED DESCRIPTION:
Over a lifetime, about half of women and a quarter of men will suffer a fragility bone fracture [1, 2], mostly due to falling [2]. Among the most serious and common fractures are hip fractures, reaching significant levels of mortality [2] and disability [3]. Hip fracture is an increasingly important problem internationally, particularly in developing countries, due to the growth in the numbers of older people. It is estimated that in 2050 the global number of hip fractures will be between 7.3 and 21.3 million [4] and the cost with the treatment will be approximately of 131.5 billion dollars [5], due the population increase.

Physical and psychological limitations post-fracture, such as decreased mobility [6] and muscle strength of lower limbs [7], deficit balance [6], lack of trust [7], fear of falling [6] and increased risk of falls [8], hamper around 40% of older people from returning to their daily activities to live independently and safely [3, 9]. Even after two years of injury, more than half of the elderly do not regain the functional level prior to injury [10], persisting with moderate to high risk of falls [6].

Risk of falls and future falls in this population may be due either to physical limitations [11, 12] (due to insufficient recovery of balance, muscle strength and consequently mobility) and the fact they have already suffered a fracture previously [13], further increasing the chances of new fractures in this population [14].

There is no consensus about the best intervention for functionality of the elderly after hip fracture. However, recently different exercise programs have been suggested to improve the mobility of these patients [8]. Some studies have shown the effectiveness of rehabilitation programs in the period of up to 6 months after injury [15-18]. Although, few studies have explored the late period rehabilitation (over 6 months) [19, 20], when functional limitations can persist due to inadequate dose as well as the type of exercise performed. Population in Brazil is growing age in one of the fastest rates in the world and will be even greater in the coming decades. The number of seniors will double between 2002 and 2020, from 15 million to 32 million and reach 64 million by 2050 (about 30% of the total population in Brazil) [21]. Furthermore, the elderly aged 80 and over will increase exponentially over the next four decades, putting a growing and disproportionate demand on the health system and social support [21].

The purpose of this study is to determine if an exercise program training for people who have suffered a fall-related hip fracture will improve functional mobility when compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* After the first hip fragility fracture following a fall from standing height or while turning
* Surgically treated in the later stage of rehabilitation phase (6 months up to 2 years after the fracture).

Exclusion Criteria:

* Sustained a hip fracture trauma due to falls from higher surfaces or motor vehicle accidents or due to a tumors or disease (other than osteoporosis)
* Several cognitive impairment, assessed by Mini-Mental State Examination adjusted for educational level [22];
* Inability to walk, either with walking aid;
* Progressive or severe neurological disease (e.g., Parkinson's disease, stroke);
* Communication disability (several uncompensated visual or hearing deficits);
* Medical condition contraindications exercise (e.g. unstable angina, severe valvular heart disease, large or expanding aortic aneurysm, etc.) [23];
* Engaged in a regular exercise program, with a frequency more or equal than twice a week, 30 minutes a day (excluding walking and senior dance) [24].

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Lower extremity function (Short Physical Performance Battery (SPPB) | Change from baseline will be assessed at 6 and 12 months
  will be measured by theSPPB [27], that consists of three blocks of tests that assess static balance, walking speed and, indirectly, the strength of the lower limbs (sitting and standing from a chair unassisted). Each test has a score of zero (worst performance) to 4 points (best performance), summing a total final score of 12 points. Change from baseline will be assessed at 6 and 12 months.

SECONDARY OUTCOMES:
Physiological risk of falls (Profile Physiological Assessment long version (PPA) | Change from baseline will be assessed at 6 and 12 months
  will be measured by the PPA [12] which provides an overall score for risk of falling through a series of tests that evaluates the systems involved in the postural stability system. The results are computed on a software specifically developed for the test that generates a report assessing the risk of falls including 4 components: the individuals score on a global chart of fall risk, profile of the individuals performance in the tests, indicating in a table individuals performance in relation to the standards of the same age. Additionally, individual score for muscle strength, reaction time test, balance, sway and coordination will be also ascertained. Change from baseline will be assessed at 6 and 12 months.
Functional performance (WHO Disability Assessment Schedule (WHODAS II) | Change from baseline will be assessed at 6 and 12 months
  measured by the WHODAS II [29]. This scale measures the population health and functionality in 6 domains: cognition, mobility, self-care, interpersonal relationships, daily activities and participation. It was developed by WHO with theoretical model to the International Classification of Functioning, Disability and Health (ICF), and it is not intended for any specific health condition. This short version assesses the difficulty degree of performing 12 activities in past 30 days, which can be classified as none, mild, moderate, severe and extreme (cannot be performed). The degree of difficulty reported is based on the presence of increased effort, discomfort or pain, slowness or the presence of some change in the way of doing the activity. Change from baseline will be assessed at 6 and 12 months.
Quality of life (WHOQOL-bref) | Change from baseline will be assessed at 6 and 12 months
  measured by WHOQOL-bref [30], consists of 26 questions divided in 4 domains: physical, psychological, social relationships and environment. The questionnaire is based on the last 2 weeks of the participant and evaluated, for example, how safe he/she feel in her/his daily life and how satisfied is he/she with his/her ability to perform daily life activities. Change from baseline will be assessed at 6 and 12 months.
Physical activity intensity (Planned Exercise Questionnaire - IPEQ_W) | Change from baseline will be assessed at 6 and 12 months
  will be measured by the IPEQ_W [31], ten questions designed to measure physical activity planned and unplanned for older people. The version estimates the intensity of physical activity during the last week will be used. The participant will be questioned for the frequency (every day, 3-6 times per week, twice a week, once a week or less than once per week) and duration of activity (less than 15 minutes per day, more than 15 minutes and under 30 minutes per day, more than 30 minutes and less than 1 hour, less over 1 h and 2 h per day more and less than 4h per day 2h, 4h, and daily or more). The total score is derived by multiplying the frequency categories by categories of activity duration, expressed in hours per week. The ICC for the IPEQ_W total score was 0.81. The concurrent validity was adequate whereas the instrument was able to identify older people of different ages and degrees of disability. Change from baseline will be assessed at 6 and 12 months.
Occurrence of falls | Change from baseline will be assessed at 6 and 12 months
  will be assessed by monthly phone calls to participants. They will be encouraged to fill the diary that containing the record daily and the number of falls. A structured questionnaire will be used to identify possible falls and their consequences. The intervention group will be compared to control group at 6 and 12 months follow-up in relation to the number of falls, the incidence of falls and the proportion of elderly fallers. Change from baseline will be assessed at 6 and 12 months.
Usual gait speed (evaluate acceleration and deceleration using a stopwatch) | Change from baseline will be assessed at 6 and 12 months
  will be evaluated on a distance of 4.6 meters, including 2 meters for acceleration and 2 meters for deceleration using a stopwatch. The participant will be instructed to walk at their normal pace as if they were going to buy something at the grocery store. The time that the elderly takes to complete the course will be recorded three times. The computed velocity in meters per second will be calculated dividing the course in meters by the time taken to complete the course. The average of three attempts will be used. The use of walking aids will be allowed during the test [28]. Change from baseline will be assessed at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Monica R Perracini, Phd, Principal Investigator — Universidade Cidade de São Paulo
Locations (1):
- Universidade Cidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Akesson K, Marsh D, Mitchell PJ, McLellan AR, Stenmark J, Pierroz DD, Kyer C, Cooper C; IOF Fracture Working Group. Capture the Fracture: a Best Practice Framework and global campaign to break the fragility fracture cycle. Osteoporos Int. 2013 Aug;24(8):2135-52. doi: 10.1007/s00198-013-2348-z. Epub 2013 Apr 16. PMID 23589162
- [Background] Johnell O, Kanis J. Epidemiology of osteoporotic fractures. Osteoporos Int. 2005 Mar;16 Suppl 2:S3-7. doi: 10.1007/s00198-004-1702-6. Epub 2004 Sep 8. PMID 15365697
- [Background] Magaziner J, Simonsick EM, Kashner TM, Hebel JR, Kenzora JE. Predictors of functional recovery one year following hospital discharge for hip fracture: a prospective study. J Gerontol. 1990 May;45(3):M101-7. doi: 10.1093/geronj/45.3.m101. PMID 2335719
- [Background] Gullberg B, Johnell O, Kanis JA. World-wide projections for hip fracture. Osteoporos Int. 1997;7(5):407-13. doi: 10.1007/pl00004148. PMID 9425497
- [Background] Johnell O. The socioeconomic burden of fractures: today and in the 21st century. Am J Med. 1997 Aug 18;103(2A):20S-25S; discussion 25S-26S. doi: 10.1016/s0002-9343(97)90023-1. PMID 9302894
- [Background] Shumway-Cook A, Ciol MA, Gruber W, Robinson C. Incidence of and risk factors for falls following hip fracture in community-dwelling older adults. Phys Ther. 2005 Jul;85(7):648-55. PMID 15982171
- [Background] Portegijs E, Edgren J, Salpakoski A, Kallinen M, Rantanen T, Alen M, Kiviranta I, Sihvonen S, Sipila S. Balance confidence was associated with mobility and balance performance in older people with fall-related hip fracture: a cross-sectional study. Arch Phys Med Rehabil. 2012 Dec;93(12):2340-6. doi: 10.1016/j.apmr.2012.05.022. Epub 2012 Jun 12. PMID 22698990
- [Background] Handoll HH, Sherrington C, Mak JC. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2011 Mar 16;(3):CD001704. doi: 10.1002/14651858.CD001704.pub4. PMID 21412873
- [Background] Rubenstein LZ. Falls in older people: epidemiology, risk factors and strategies for prevention. Age Ageing. 2006 Sep;35 Suppl 2:ii37-ii41. doi: 10.1093/ageing/afl084. PMID 16926202
- [Background] Magaziner J, Hawkes W, Hebel JR, Zimmerman SI, Fox KM, Dolan M, Felsenthal G, Kenzora J. Recovery from hip fracture in eight areas of function. J Gerontol A Biol Sci Med Sci. 2000 Sep;55(9):M498-507. doi: 10.1093/gerona/55.9.m498. PMID 10995047
- [Background] Sherrington C, Tiedemann A, Cameron I. Physical exercise after hip fracture: an evidence overview. Eur J Phys Rehabil Med. 2011 Jun;47(2):297-307. Epub 2011 May 10. PMID 21555983
- [Background] Lord SR, Menz HB, Tiedemann A. A physiological profile approach to falls risk assessment and prevention. Phys Ther. 2003 Mar;83(3):237-52. PMID 12620088
- [Background] Perracini MR, Ramos LR. [Fall-related factors in a cohort of elderly community residents]. Rev Saude Publica. 2002 Dec;36(6):709-16. doi: 10.1590/s0034-89102002000700008. Portuguese. PMID 12488937
- [Background] Berry SD, Samelson EJ, Hannan MT, McLean RR, Lu M, Cupples LA, Shaffer ML, Beiser AL, Kelly-Hayes M, Kiel DP. Second hip fracture in older men and women: the Framingham Study. Arch Intern Med. 2007 Oct 8;167(18):1971-6. doi: 10.1001/archinte.167.18.1971. PMID 17923597
- [Background] Binder EF, Brown M, Sinacore DR, Steger-May K, Yarasheski KE, Schechtman KB. Effects of extended outpatient rehabilitation after hip fracture: a randomized controlled trial. JAMA. 2004 Aug 18;292(7):837-46. doi: 10.1001/jama.292.7.837. PMID 15315998
- [Background] Mangione KK, Palombaro KM. Exercise prescription for a patient 3 months after hip fracture. Phys Ther. 2005 Jul;85(7):676-87. PMID 15982174
- [Background] Sherrington C, Lord SR, Herbert RD. A randomised trial of weight-bearing versus non-weight-bearing exercise for improving physical ability in inpatients after hip fracture. Aust J Physiother. 2003;49(1):15-22. doi: 10.1016/s0004-9514(14)60184-7. PMID 12600250
- [Background] Mitchell SL, Stott DJ, Martin BJ, Grant SJ. Randomized controlled trial of quadriceps training after proximal femoral fracture. Clin Rehabil. 2001 Jun;15(3):282-90. doi: 10.1191/026921501676849095. PMID 11386398
- [Background] Sherrington C, Lord SR, Herbert RD. A randomized controlled trial of weight-bearing versus non-weight-bearing exercise for improving physical ability after usual care for hip fracture. Arch Phys Med Rehabil. 2004 May;85(5):710-6. doi: 10.1016/s0003-9993(03)00620-8. PMID 15129393
- [Background] Sherrington C, Lord SR. Home exercise to improve strength and walking velocity after hip fracture: a randomized controlled trial. Arch Phys Med Rehabil. 1997 Feb;78(2):208-12. doi: 10.1016/s0003-9993(97)90265-3. PMID 9041904
- [Background] Gragnolati M, Jorgensen OH, Rocha R, Fruttero A. Growing Old in an Older Brazil: Implicatios of population aging on growth, porverty, public finance, and service delivery. Washington, D.C.: The World Bank; 2011.
- [Background] Bertolucci PH, Brucki SM, Campacci SR, Juliano Y. [The Mini-Mental State Examination in a general population: impact of educational status]. Arq Neuropsiquiatr. 1994 Mar;52(1):1-7. Portuguese. PMID 8002795
- [Background] Frankel JE, Bean JF, Frontera WR. Exercise in the elderly: research and clinical practice. Clin Geriatr Med. 2006 May;22(2):239-56; vii. doi: 10.1016/j.cger.2005.12.002. PMID 16627076
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1435-45. doi: 10.1249/mss.0b013e3180616aa2. PMID 17762378
- [Background] Singh MA. Exercise comes of age: rationale and recommendations for a geriatric exercise prescription. J Gerontol A Biol Sci Med Sci. 2002 May;57(5):M262-82. doi: 10.1093/gerona/57.5.m262. No abstract available. PMID 11983720
- [Background] Freire AN, Guerra RO, Alvarado B, Guralnik JM, Zunzunegui MV. Validity and reliability of the short physical performance battery in two diverse older adult populations in Quebec and Brazil. J Aging Health. 2012 Aug;24(5):863-78. doi: 10.1177/0898264312438551. Epub 2012 Mar 15. PMID 22422762
- [Background] Fleck MP, Louzada S, Xavier M, Chachamovich E, Vieira G, Santos L, Pinzon V. [Application of the Portuguese version of the abbreviated instrument of quality life WHOQOL-bref]. Rev Saude Publica. 2000 Apr;34(2):178-83. doi: 10.1590/s0034-89102000000200012. Portuguese. PMID 10881154
- [Background] Ustun TB, Chatterji S, Kostanjsek N, Rehm J, Kennedy C, Epping-Jordan J, Saxena S, von Korff M, Pull C; WHO/NIH Joint Project. Developing the World Health Organization Disability Assessment Schedule 2.0. Bull World Health Organ. 2010 Nov 1;88(11):815-23. doi: 10.2471/BLT.09.067231. Epub 2010 May 20. PMID 21076562
- [Background] Merom D, Delbaere K, Cumming R, Voukelatos A, Rissel C, Van Der Ploeg HP, Lord SR. Incidental and Planned Exercise Questionnaire for seniors: validity and responsiveness. Med Sci Sports Exerc. 2014;46(5):947-54. doi: 10.1249/MSS.0000000000000196. PMID 24743107
- [Background] Ruggero CR, Bilton TL, Teixeira LF, Ramos Jde L, Alouche SR, Dias RC, Perracini MR. Gait speed correlates in a multiracial population of community-dwelling older adults living in Brazil: a cross-sectional population-based study. BMC Public Health. 2013 Feb 28;13:182. doi: 10.1186/1471-2458-13-182. PMID 23448191
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134
- [Derived] Lima CA, Sherrington C, Guaraldo A, Moraes SA, Varanda RD, Melo JA, Kojima KE, Perracini M. Effectiveness of a physical exercise intervention program in improving functional mobility in older adults after hip fracture in later stage rehabilitation: protocol of a randomized clinical trial (REATIVE Study). BMC Geriatr. 2016 Nov 29;16(1):198. doi: 10.1186/s12877-016-0370-7. PMID 27894271